CLINICAL TRIAL: NCT05333731
Title: To Study the Effectiveness and Safety of Oxytocin Induction in Full Term Pregnant Women With Cesarean Section of Prelabor Rupture of Membranes: a Multi-center, Prospective, Observational Study
Brief Title: Oxytocin Induction in Full Term Pregnant Women With Cesarean Section of Prelabor Rupture of Membranes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: JPPTOLAC-02
Record Dates: First submitted 2022-02-08; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Failed Trial of Labor, Unspecified, With Delivery; Failed VBAC (Vaginal Birth After Caesarean); Prelabor Rupture of Membranes; Failed Induction (of Labor) by Oxytocin
MeSH Terms: conditions — Fetal Membranes, Premature Rupture | interventions — Oxytocin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cesarean section group: In the cesarean section group, all the pregnant women had only one prior cesarean section.
  Interventions: Drug: Oxytocin
- Non-cesarean section group: In the non-cesarean section group, all the pregnant women are primipara, and never had a cesarean section.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — In the two groups, if spontaneous labor does not occur after PROM, they all receive the oxytocin for up to 24h.

SUMMARY:
This study is a multi-center, prospective, observational clinical trial study. 528 full-term pregnant women will be enrolled as subjects, and the ratio of eligible subjects in the two groups is 1:1. In the cesarean section group, full term pregnant women with prelabor rupture of membrane (PROM) who are willing to try the trial of labor after cesarean (TOLAC) and in accordance with the criteria according to the 2016 China vaginal birth after cesarean (VBAC) clinical management guidelines will be enrolled and recorded by our homemade registration form of TOLAC. In the non-cesarean section group, pregnant women after 37 weeks of gestation with PROM but without vaginal labor contraindications will be enrolled. Whether in the cesarean section group or non-cesarean section group, if spontaneous labor does not occur, and they all will be induced by oxytocin. After 24 hours, their final delivery mode will be recorded. In the following 42 days postpartum, their complications and the neonatal outcome will be followed up.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers sign the informed consent;
2. Age: 20-40 years;
3. Singleton, a cephalic presentation;
4. No contradiction to vaginal delivery;
5. gestation: 37~42 weeks;
6. With prelabor rupture of membrane.

Exclusion criteria:

1. Konwn contraindication to vaginal delivery or severe complications;
2. Multiple gestation;
3. Uterine malformation;
4. Severe psychiatric disorder;
5. Without family's support.

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: In the cesarean section group, the extra inclusion criteria includes:
  Only one prior low transverse uterine incision;
  Extra exclusion criteria:
  1. With mutiple history of c esction;
  2. Prior extensive transfundal uterine surgery, such as for fetal surgery, myomectomy, or uterine reconstruction; Prior classical vertical uterine incision, or an inverted "T" or "J" incision;
  3. Short interpregnancy interval;
  4. Prior uterine rupture or dehiscence, or cesarean scar pregnancy;
  5. Evaluated fetal birth weight> 4000 g.
  In the non-cesarean section group, the extra criteria should include:
  nulliparous
Sampling Method: Probability Sample
Enrollment: 528 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Vignial birth rate | 24 hours
  After the treatment of oxytocin induction for up tp 24 hours, the mode of delivery will be konwn and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Prelabor Rupture of Membranes: ACOG Practice Bulletin, Number 217. Obstet Gynecol. 2020 Mar;135(3):e80-e97. doi: 10.1097/AOG.0000000000003700. PMID 32080050
- [Background] Bellussi F, Livi A, Diglio J, Lenzi J, Magnani L, Pilu G. Timing of induction for term prelabor rupture of membranes and intravenous antibiotics. Am J Obstet Gynecol MFM. 2021 Jan;3(1):100245. doi: 10.1016/j.ajogmf.2020.100245. Epub 2020 Oct 6. PMID 33451610
- [Background] Fishel Bartal M, Sibai BM, Ilan H, Fried M, Rahav R, Alexandroni H, Schushan Eisan I, Hendler I. Trial of labor after cesarean (TOLAC) in women with premature rupture of membranes. J Matern Fetal Neonatal Med. 2020 Sep;33(17):2976-2982. doi: 10.1080/14767058.2019.1566312. Epub 2019 Jan 17. PMID 30652525
- [Background] Middleton P, Shepherd E, Flenady V, McBain RD, Crowther CA. Planned early birth versus expectant management (waiting) for prelabour rupture of membranes at term (37 weeks or more). Cochrane Database Syst Rev. 2017 Jan 4;1(1):CD005302. doi: 10.1002/14651858.CD005302.pub3. PMID 28050900